CLINICAL TRIAL: NCT04053127
Title: Respiratory-Gated Vagal Nerve Stimulation for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Robert Edwards, Clinical Psychologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RAVANS_PILOT
Record Dates: First submitted 2018-10-02; First posted 2019-08-12 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Chronic Pain
Keywords: vagus nerve stimulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RAVANS (Experimental): Electrodes will be placed in the auricle of the left ear. Electrical stimulation to these electrodes will be provided by a current-constant stimulator (Urostim, Schwa-Medico). Stimulation will be gated, with 1-second delay, after peak inhalation (i.e. during exhalation). Respiratory gating for stimulation will require real-time evaluation of the respiratory cycle. The study will use a belt system constructed in-house, and similar to the system used in several previous studies. A pneumatic belt will be placed around the subject's lower thorax. Once electrodes are set up, subjects will be asked to rate stimulation intensity on a NRS of 0 to 10 (0: no sensation, 10: pain detection threshold). Current intensity will be set to achieve moderate to strong (but not painful) sensation, and this current intensity will be used on subsequent stimulation runs.
  Interventions: Device: RAVANS
- non-RAVANS (Sham Comparator): For sessions randomized to sham stimulation, the electrodes in the ear will remain as described above, but the leads will be disconnected from the stimulator. Subjects will be instructed that for this session they may or may not feel pulsing in their ear, and that the goal is to ensure that the stimulus was not painful.
  Interventions: Device: RAVANS

INTERVENTIONS:
Device: RAVANS — Electrical stimulation of somatosensory vagal afferent receptors in the ear modulated by respiration.
  Other Names: Respiratory-gated Auricular Vagal Afferent Nerve Stimulation

SUMMARY:
Vagus Nerve Stimulation (VNS) is a validated and FDA-approved therapy that has improved the lives of many individuals with epilepsy and depression and has shown promise for treating chronic pain. However, there is moderate morbidity associated with the surgical procedure and maintenance of VNS. The study team has developed a novel, non-invasive procedure based on the neurobiology of VNS treatment which is termed Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS). The investigators hope to maximize efficacy and better understand applicability of RAVANS by applying this to chronic pain patients with a range of psychiatric and psychological comorbidity. This high-distress subpopulation of chronic pain patients has been notoriously difficult to treat and is in need of new, innovative therapies. The investigators propose applying electrical stimulation of the somatosensory vagal afferent receptors in the ear using transcutaneous-VNS (t-VNS) during the exhalation phase of breathing in order to augment the clinical efficacy of t-VNS.

This proposal includes a single blinded, controlled design for testing the impact of RAVANS therapy on pain and mood fro chronic pain. Patients will complete 2 in-person visits, one with RAVANS therapy and one with non-RAVANS stimulation. During each session, participants will complete questionnaires, quantitative sensory testing (QST), and receive either real or sham RAVANS stimulation.

DETAILED DESCRIPTION:
Testing will occur over the course of 2 2-3 hour study visits. After completing consent forms, participants will complete questionnaires and undergo baseline Quantitative Sensory Testing (QST). After baseline sensory testing and completion of measures, participants will complete a 30-minute rest period during which time they are instructed to relax and regulate their breathing. After the rest, they will receive a 30-minute RAVANS or non-RAVANS stimulation. Following the RAVANS stimulation, participants will again undergo QST testing. Throughout the session, subjects will rate pain and mood using numeric rating scales and physiological monitoring will occur as described below.

RAVANS stimulation Electrodes will be placed in the auricle of the left ear. Electrical stimulation to these electrodes will be provided by a current-constant stimulator (Urostim, Schwa-Medico). Stimulation will be gated, with 1-second delay, after peak inhalation (i.e. during exhalation). Respiratory gating for stimulation will require real-time evaluation of the respiratory cycle. The study will use a belt system constructed in-house, and similar to the system used in several previous studies. A pneumatic belt will be placed around the subject's lower thorax. Once electrodes are set up, subjects will be asked to rate stimulation intensity on a NRS of 0 to 10 (0: no sensation, 10: pain detection threshold). Current intensity will be set to achieve moderate to strong (but not painful) sensation, and this current intensity will be used on subsequent stimulation runs.

Non-RAVANS stimulation For sessions randomized to sham stimulation, the electrodes in the ear will remain as described above, but the leads will be disconnected from the stimulator. Subjects will be instructed that for this session they may or may not feel pulsing in their ear, and that the goal is to ensure that the stimulus was not painful.

Physiological Monitoring In addition to respiration, which by necessity will be monitored with the pneumatic belt as part of the RAVANS procedure, the investigators will also collect ECG data. The ECG signal will also be acquired by a laptop device system, temporally locked to the respiratory signal. The ECG can be used to quantify heart rate and heart rate variability.

Sensory Tests to be Completed at Baseline and After Experimental Condition:

These procedures are similar to those used in ongoing QST studies (e.g., IRB protocols 2009P001020, 2010P000978, 2015P002373).

Mechanical pain: Responses to punctate mechanical stimuli will be measured using a standard set of weighted probes that provide estimates of pain threshold and mechanical temporal summation. Series of 10 stimuli (with 1-second inter-stimulus intervals) will be used to assess the temporal summation of pain that occurs with rapid administration of identical stimuli. A Somedic pressure algometer will be utilized to assess responses to pressure stimulation at several anatomical sites. Pain pressure thresholds (PPT) will be determined twice at the knee, trapezius, and thumb. Mechanical pressure will be applied using a 0.5-cm2 probe covered with 1mm polypropylene pressure-transducing material; pressure is increased at a steady rate of 30 kPA/s until the subject indicates that the pressure has become painful. Finally, the study will use cuff algometry to assess responses to sustained mechanical pressure. A Hokanson rapid cuff inflator will be used to inflate a standard blood pressure cuff around the gastrocnemius muscle to a moderately painful level for up to 2 minutes. Participants will indicate when the pressure first becomes painful (i.e., pain threshold) and will provide pain ratings every 30 seconds. As with each of these psychophysical testing procedures, participants are informed that they may terminate the procedure at any time.

ELIGIBILITY:
Inclusion Criteria:

1. age 21-65.
2. chronic pain lasting for more than 6 months as the primary complaint.
3. typical pain ratings ≥ 3/10 on a visual analogue scale.
4. able to speak and understand English.

Exclusion Criteria:

1. evidence of delirium, dementia, psychosis, or other cognitive impairment preventing completion of study procedures.
2. history of cardiac or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome.
3. current peripheral neuropathy.
4. current pregnancy, or intention to become pregnant during the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Mechanical Temporal Summation | immediately post-RAVANS stimulation
  Increases in pain with repeated mechanical stimulation
Pressure Pain Sensitivity | immediately post-RAVANS stimulation
  Thresholds for pressure pain assessed at several body sites

SECONDARY OUTCOMES:
Pain Severity | immediately post-RAVANS
  Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Napadow, Ph.D., Principal Investigator — MGH & BWH
Locations (1):
- Robert Edwards, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared.